CLINICAL TRIAL: NCT05174065
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Apremilast (AMG 407) in Japanese Subjects With Palmoplantar Pustulosis (PPP)
Brief Title: Phase 3, Randomized Study of Apremilast in Japanese Participants With Palmoplantar Pustulosis (PPP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20200195
Record Dates: First submitted 2021-12-14; First posted 2021-12-30 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-02

CONDITIONS: Palmoplantar Pustulosis
Keywords: Palmoplantar Pustulosis; PPP; AMG 407; Apremilast; Otezla
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Apremilast (Experimental): Apremilast will be administered to participants twice daily (BID)
  Interventions: Drug: Apremilast
- Placebo and Apremilast (Experimental): Matching placebo will be administered to participants twice daily (BID) until week 16. After week 16, Apremilast will be administered to participants BID.
  Interventions: Drug: Apremilast; Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Oral tablets
  Other Names: Otezla; AMG 407
Drug: Placebo — Oral tablets
  Arms: Placebo and Apremilast

SUMMARY:
The primary objective of the study is to evaluate the efficacy of apremilast (AMG 407) twice daily (BID) compared with placebo in participants with Palmoplantar Pustulosis (PPP).

ELIGIBILITY:
* Key Inclusion Criteria

  * Japanese participants ≥ 18 years of age upon entry into initial screening
  * Palmoplantar pustulosis diagnosis with or without pustulotic arthro-osteitis (PAO) for no less than 24 weeks
  * PPPASI total score of ≥12 at screening and at baseline
  * Moderate or severe pustules/vesicles on palms or soles (PPPASI severity score ≥2) at screening and at baseline
  * Inadequate response (defined as repeated relapsing-remitting in the same location for a 24-week period) to topical treatments prior to or at screening
* Key Exclusion Criteria

  * Changes in disease severity during screening (PPPASI total score change ≥ 5 improvement, from screening to baseline)
  * Periodontitis requiring treatment
  * Chronic or recurrent tonsillitis or sinusitis requiring any continuous treatment
  * Has a diagnosis of plaque-type psoriasis at baseline
  * Has the presence of pustular psoriasis on any part of the body other than the palms and soles
  * Has evidence of skin conditions of hand and feet at baseline that would interfere with evaluations of the effect of Investigational Product
  * Has unstable cardiovascular disease, defined as a recent clinical deterioration or a cardiac hospitalization within 12 weeks prior to screening
  * Malignancy or history of malignancy
  * Participant has received any procedures for focal infection within 24 weeks of baseline
  * Female participants who are breastfeeding or who plan to breastfeed while on study
  * Female participants of childbearing potential with a positive pregnancy test
  * Had prior treatment with apremilast
  * Has a prior medical history of suicide attempt at any time in the participant's lifetime prior to signing of informed consent or randomization, or major psychiatric illness requiring hospitalization within the last 3 years prior to signing of informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (40):
- Japan (40):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Toho University Sakura Medical Center, Sakura-shi, Chiba
  - Ehime University Hospital, Toon-shi, Ehime
  - Kusuhara Dermatology Clinic, Fukuoka, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Higuchi Dermatology Urology Clinic, Kasuga-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Nagata Dermatology Clinic, Ogori-shi, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Central Japan International Medical Center, Minokamo-shi, Gifu
  - Motomachi Dermatology Clinic, Asahikawa-shi, Hokkaido
  - Asahikawa Medical University Hospital, Asahikawa-shi, Hokkaido
  - Medical corporation kojinkai Chitose dermatology and plastic surgery clinic, Chitose-shi, Hokkaido
  - Shinoro Dermatology Clinic, Sapporo, Hokkaido
  - Medical Corporation Kojinkai Kitago Dermatology Clinic, Sapporo, Hokkaido
  - Shibaki Dermatology Clinic, Sapporo, Hokkaido
  - Medical Corporation Kojinkai Sapporo Skin Clinic, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Nomura Dermatology Clinic, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nankoku-shi, Kochi
  - Nagaoka Red Cross Hospital, Nagaoka-shi, Niigata
  - Oita University Hospital, Yufu-shi, Oita Prefecture
  - Nippon Life Hospital, Osaka, Osaka
  - Medical Corporation Goto Dermatology Clinic, Osaka, Osaka
  - Dermatology and Ophthalmology Kume Clinic, Sakai-shi, Osaka
  - Yoshikawa Skin Clinic, Takatsuki-shi, Osaka
  - Dokkyo Medical University Saitama Medical Center, Koshigaya-shi, Saitama
  - Pansy Skin Clinic, Saitama-shi, Saitama
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Tokyo Teishin Hospital, Chiyoda-ku, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Seibo International Catholic Hospital, Shinjuku-ku, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Terui T, Okubo Y, Kobayashi S, Morita A, Imafuku S, Tada Y, Abe M, Strober B, Gooderham M, Zhang W, Shimauchi J, Yaguchi M, Kimura T, Ogawa R, Amouzadeh H, Murakami M. Apremilast in Japanese patients with palmoplantar pustulosis: A randomized, Phase 3 trial. J Eur Acad Dermatol Venereol. 2025 Nov 26. doi: 10.1111/jdv.70166. Online ahead of print. PMID 41297955
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with palmoplantar pustulosis (PPP) took part in the study at 40 centers in Japan between 08 March 2022 and 01 June 2024.
Pre-assignment Details: A total of 176 participants were enrolled in the placebo-controlled period. Of these, 172 participants were enrolled in the active treatment period.
Groups:
- Placebo-controlled Period: Placebo: Participants took oral placebo matching apremilast tablets twice daily (BID) from Week 0 to Week 16 during the placebo-controlled period.
- Placebo-controlled Period: Apremilast: Participants took oral apremilast tablets BID, starting at a dose of 10 mg and gradually increasing to the target 30 mg dose over 5 days, from Week 0 to Week 16 during the placebo-controlled period.
- Active Treatment Period: Apremilast: Participants who were randomized to placebo during the placebo-controlled period took oral apremilast tablets BID, starting at a dose of 10 mg and gradually increasing to the target 30 mg dose over 5 days, from Week 16 to Week 52. Participants who were randomized to apremilast during the placebo-controlled period took oral 30 mg apremilast tablets BID from Week 16 to Week 52.
Period: Placebo-controlled Period
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Apremilast | Active Treatment Period: Apremilast
Started | 88 | 88 | 0 (This arm was included in the active treatment period only.)
Received Apremilast or Placebo During Placebo-controlled Period | 88 | 88 | 0
Completed (Completed investigational product treatment in the placebo-controlled period.) | 86 | 86 | 0
Not Completed | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Other | 0 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0
Period: Apremilast Active Treatment Period
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Apremilast | Active Treatment Period: Apremilast
Started | 0 (This arm was included for the placebo-controlled period.) | 0 (This arm was included for the placebo-controlled period.) | 172
Received Apremilast During the Active Treatment Period | 0 | 0 | 172
Completed | 0 | 0 | 164
Not Completed | 0 | 0 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat Population: Included all randomized participants (i.e., participants who entered the placebo-controlled period).
Groups:
- Placebo-controlled Period: Placebo: Participants took oral placebo matching apremilast tablets BID from Week 0 to Week 16.
- Placebo-controlled Period: Apremilast: Participants took oral apremilast tablets BID, starting at a dose of 10 mg and gradually increasing to the target 30 mg dose over 5 days, from Week 0 to Week 16.
- Total: Total of all reporting groups
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Apremilast | Total
Number analyzed (Participants) | 88 | 88 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (11.35) | 57.0 (11.32) | 56.5 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 69 | 141
  Male | 16 | 19 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 88 | 88 | 176
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 88 | 88 | 176

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved at Least a 50% Reduction From Baseline in Palmoplantar Pustulosis Area and Severity Index (PPPASI) Total Score (PPPASI-50) at Week 16
Description: A PPPASI 50 response is defined as a ≥ 50% reduction in PPPASI total score from baseline.
  The PPPASI is a system used for assessing and grading the severity (in terms of erythema, pustules/vesicle and desquamation/scale) and area of PPP lesions and their response to therapy. The PPPASI produces a numeric score that can range from 0 to 72, with a higher score indicating more severe disease.
  Participants who discontinued investigational product before week 16 due to lack of efficacy, adverse event, or use of protocol-prohibited medication (intercurrent events) were to be considered as treatment failures as the result of the intercurrent event and the PPPASI-50 values for visits on and after the intercurrent event were imputed as non-responders. The missing PPPASI-50 values due to the other reasons were imputed using the multiple imputation method.
Time Frame: Baseline and Week 16
Population: ITT Population: Included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Apremilast
Number analyzed (Participants) | 88 | 88
percentage of participants | 35.3 [25.3 to 45.4] | 67.8 [57.9 to 77.6]
Statistical Analysis 1: Comparison: Placebo-controlled Period: Placebo vs Placebo-controlled Period: Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted for the stratification factors of rounded PPPASI total score range (≤ 20/21 to 30/≥ 31) and focal infection status (yes/no) at baseline; Adjusted Difference in Proportion = 32.6, 95% CI 2-sided [18.7 to 46.5] — Based on the Cochran-Mantel-Haenszel method adjusting for the stratification factors. The adjusted difference in proportion was the weighted average of the treatment differences across strata

2. Secondary Outcome: Change From Baseline in PPPASI Total Score at Week 16
Description: The PPPASI is a system used for assessing and grading the severity (in terms of erythema, pustules/vesicle and desquamation/scale) and area of PPP lesions and their response to therapy. The PPPASI produces a numeric score that can range from 0 to 72, with a higher score indicating more severe disease. A negative change from baseline indicates a reduction in disease severity.
  The continuous endpoints collected on and after the participant experienced treatment failure as the result of intercurrent event (IE) (investigational product discontinuation due to lack of efficacy, adverse event, or protocol-prohibited medication use), the baseline value of corresponding endpoint were assigned to the data on and after IE up to Week 16 regardless of the observed data. The missing data due to other reasons will not be imputed considering the mixed-effects model for repeated measures (MMRM) application.
Time Frame: Baseline and Week 16
Population: ITT Population: Included all randomized participants. Only participants with observed data, including participants who had intercurrent events and were assigned baseline values were included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Apremilast
Number analyzed (Participants) | 86 | 87
score on a scale | -5.98 (0.999) | -12.12 (1.002)
Statistical Analysis 1: Comparison: Placebo-controlled Period: Placebo vs Placebo-controlled Period: Apremilast; Test type: Superiority; p < 0.0001, MMRM; With treatment group, visit time, treatment-by-time interaction, and stratification factors as fixed effect, and the baseline value as a covariate; Difference in Least Squares Mean = -6.13, 95% CI 2-sided [-8.57 to -3.69] — Apremilast - Placebo

3. Secondary Outcome: Change From Baseline in Palmoplantar Pustulosis Severity Index (PPSI) Total Score at Week 16
Description: The PPSI is a system used for assessing and grading the severity of PPP lesions and their response to therapy. Evaluation of skin lesion site are assessed separately for erythema, pustules/vesicle and desquamation/scale, where each are rated on a scale of 0 to 4 and summed to produce a numeric total score than can range from 0 to 12, with a higher score indicating more severe disease. A negative change from baseline indicates a reduction in disease severity.
  The continuous endpoints collected on and after the participant experienced treatment failure as the result of IE (investigational product discontinuation due to lack of efficacy, adverse event, or protocol-prohibited medication use), the baseline value of corresponding endpoint were assigned to the data on and after IE up to Week 16 regardless of the observed data. The missing data due to other reasons will not be imputed considering the MMRM application.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Apremilast
Number analyzed (Participants) | 86 | 87
score on a scale | -1.9 (0.24) | -3.4 (0.24)
Statistical Analysis 1: Comparison: Placebo-controlled Period: Placebo vs Placebo-controlled Period: Apremilast; Test type: Superiority; p < 0.0001, MMRM; With treatment group, visit time, treatment-by-time interaction, and stratification factors as fixed effect, and baseline value as covariate; Difference in Least Squares Mean = -1.5, 95% CI 2-sided [-2.2 to -0.9] — Apremilast - Placebo

4. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Assessment for PPP Symptoms (Pruritus) at Week 16
Description: Participants assessed the degree of pruritus itching symptoms on palms and soles caused by PPP on a VAS. The VAS score ranged from 0 to 100. The left-hand boundary (0) on the VAS represents no itch and the right-hand boundary (100) represents itch as severe as can be imagined by the participant. A negative change from baseline indicates a reduction in disease severity.
  The continuous endpoints collected on and after the participant experienced treatment failure as the result of IE (investigational product discontinuation due to lack of efficacy, adverse event, or protocol-prohibited medication use), the baseline value of corresponding endpoint were assigned to the data on and after IE up to Week 16 regardless of the observed data. The missing data due to other reasons will not be imputed considering the MMRM application.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Apremilast
Number analyzed (Participants) | 86 | 87
score on a scale | -9.9 (2.68) | -17.6 (2.67)
Statistical Analysis 1: Comparison: Placebo-controlled Period: Placebo vs Placebo-controlled Period: Apremilast; Test type: Superiority; p = 0.0330, MMRM; [statistical method as in outcome 2, analysis 1]; Difference in Least Squares Mean = -7.8, 95% CI 2-sided [-14.9 to -0.6] — Apremilast - Placebo

5. Secondary Outcome: Change From Baseline in VAS Assessment for PPP Symptoms (Pain/Discomfort) at Week 16
Description: Participants assessed the degree of pain/discomfort symptoms on palms and soles caused by PPP on a VAS. The VAS score ranged from 0 to 100. The left-hand boundary (0) on the VAS represents no pain/discomfort and the right-hand boundary (100) represents pain/discomfort as severe as can be imagined by the participant. A negative change from baseline indicates a reduction in disease severity.
  The continuous endpoints collected on and after the participant experienced treatment failure as the result of IE (investigational product discontinuation due to lack of efficacy, adverse event, or protocol-prohibited medication use), the baseline value of corresponding endpoint were assigned to the data on and after IE up to Week 16 regardless of the observed data. The missing data due to other reasons will not be imputed considering the MMRM application.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Apremilast
Number analyzed (Participants) | 86 | 87
score on a scale | -7.5 (2.97) | -18.3 (2.96)
Statistical Analysis 1: Comparison: Placebo-controlled Period: Placebo vs Placebo-controlled Period: Apremilast; Test type: Superiority; p = 0.0076, MMRM; [statistical method as in outcome 2, analysis 1]; Difference in Least Squares Mean = -10.8, 95% CI 2-sided [-18.6 to -2.9] — Apremilast - Placebo

6. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 16
Description: The DLQI is a skin disease-specific Quality of Life (QoL) questionnaire comprised of 10 items assessing the participant's status over the previous week. The DLQI was used to assess 6 different aspects that may affect QoL: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The DLQI produces a numeric score ranging from 0 to 30, with a higher score indicating more severe disease. A negative change from baseline indicates a reduction in disease severity.
  The continuous endpoints collected on and after the participant experienced treatment failure as the result of IE (investigational product discontinuation due to lack of efficacy, adverse event, or protocol-prohibited medication use), the baseline value of corresponding endpoint were assigned to the data on and after IE up to Week 16 regardless of the observed data. The missing data due to other reasons will not be imputed considering the MMRM application.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Apremilast
Number analyzed (Participants) | 87 | 87
score on a scale | -0.8 (0.37) | -2.3 (0.37)
Statistical Analysis 1: Comparison: Placebo-controlled Period: Placebo vs Placebo-controlled Period: Apremilast; Test type: Superiority; p = 0.0036, MMRM; [statistical method as in outcome 2, analysis 1]; Difference in Least Squares Mean = -1.4, 95% CI 2-sided [-2.4 to -0.5] — Apremilast - Placebo

7. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: TEAEs were defined as any untoward medical occurrence in a participant irrespective of a causal relationship with the study treatment that began or worsened on or after the first dose of study treatment.
  A serious TEAE met at least 1 of the following criteria:
  * Resulted in death.
  * Was immediately life-threatening.
  * Required in-patient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent or significant disability/incapacity.
  * Was a congenital anomaly/birth defect.
  * Was any other medically important serious event.
  TEAEs of interest were defined as any of the following:
  * Depression.
  * Serious infection.
  * Risk of triggering suicide.
  * Serious diarrhea, nausea and vomiting.
  * Malignancies.
  * Vasculitis and Vasculopathy.
  * Serious Hypersensitivity.
  * Weight change (weight decrease).
  Clinically significant changes in body weight, vital signs and laboratory abnormalities were also recorded as TEAEs.
Time Frame: Placebo-controlled period: Day 1 to Week 16; Apremilast exposure period : Apremilast Day 1 to a maximum of Week 52 (plus 4 weeks safety follow-up)
Population: Safety Population: Included all randomized participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Apremilast Exposure Period: Apremilast: Participants who received any apremilast during the placebo-controlled or active treatment periods.
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Apremilast | Apremilast Exposure Period: Apremilast
Number analyzed (Participants) | 88 | 88 | 174
Participants
  Any TEAEs | 43 | 63 | 148
  Serious TEAEs | 1 | 1 | 9
  TEAEs of Interest | 3 | 1 | 8

ADVERSE EVENTS:
Time Frame: Placebo-controlled period: Day 1 to Week 16; Apremilast exposure period : Apremilast Day 1 to a maximum of Week 52 (plus 4 weeks safety follow-up)
Description: Safety Population: Included all randomized participants who received at least 1 dose of investigational product.
Arm/Group | Placebo-controlled Period: Placebo | Placebo-controlled Period: Apremilast | Apremilast Exposure Period: Apremilast
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/88 | 0/174
Serious Adverse Events (participants affected / at risk) | 1/88 | 1/88 | 9/174
Other Adverse Events (participants affected / at risk) | 25/88 | 46/88 | 99/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Period: Placebo (N=88) | Placebo-controlled Period: Apremilast (N=88) | Apremilast Exposure Period: Apremilast (N=174)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 2
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Pseudoaneurysm infection (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Period: Placebo (N=88) | Placebo-controlled Period: Apremilast (N=88) | Apremilast Exposure Period: Apremilast (N=174)
Diarrhoea (Gastrointestinal disorders) | 3 | 17 | 31
Faeces soft (Gastrointestinal disorders) | 1 | 15 | 22
Nausea (Gastrointestinal disorders) | 1 | 10 | 23
COVID-19 (Infections and infestations) | 4 | 4 | 18
Nasopharyngitis (Infections and infestations) | 8 | 4 | 28
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 5
Headache (Nervous system disorders) | 2 | 10 | 19
Eczema (Skin and subcutaneous tissue disorders) | 3 | 5 | 11
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 5 | 4 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT05174065/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT05174065/SAP_001.pdf